CLINICAL TRIAL: NCT03862313
Title: Assessing Repetitive Transorbital Alternating Current Stimulation in Acute Autoimmune Inflammatory Optic Neuritis Using the NextWave® 1.1 System: A Prospective, Randomized, Patient-blinded, Sham-controlled Pilot Study
Brief Title: Repetitive Transorbital Alternating Current Stimulation in Acute Autoimmune Optic Neuritis
Acronym: ACSON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primarily due to insufficient recruitment (n = 2 instead of n = 30), the study was prematurely discontinued for feasibility reasons. Neither any meaningful results on safety nor on efficacy can be reported.
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other); Swiss MS Society (Unknown); Data Management, Clinical Trials Center, Zurich, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201802353
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Acute Autoimmune Inflammatory Optic Neuritis
Keywords: optic neuritis; multiple sclerosis; repetitive transorbital alternating current stimulation; optical coherence tomography; low-contrast visual acuity
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active-rtACS arm (Experimental): Active rtACS on 10 consecutive working days, in addition to standard-of-care corticosteroid treatment.
  Interventions: Device: active-rtACS treatment
- sham-rtACS arm (Sham Comparator): Sham rtACS on 10 consecutive working days, in addition to standard-of-care corticosteroid treatment.
  Interventions: Device: sham-rtACS treatment

INTERVENTIONS:
Device: active-rtACS treatment — For the active-rtACS treatment arm, a CE-certificated proprietary class IIa medical device will be used to apply transorbital symmetrical rectangular current pulses in bursts (NextWave® 1.1 system; EBS Technologies GmbH, Germany). The stimulation protocol will be patient-individualized, with a stimulation current strength of 125% of the phosphene threshold recorded during 5Hz stimulation and stimulation frequencies between the individual's EEG alpha frequency and their flicker fusion frequency.
  Other Names: NextWave® 1.1 system, EBS Technologies GmbH, Germany
  Arms: active-rtACS arm
Device: sham-rtACS treatment — For the sham-rtACS treatment arm, exactly the same medical device, setup, time schedule, etc. will be used as for the patients of the active-rtACS arm. However, sham-treated patients will receive no actual current stimulation during the therapy sessions.
  Other Names: NextWave® 1.1 system, EBS Technologies GmbH, Germany
  Arms: sham-rtACS arm

SUMMARY:
Optic neuritis (ON) is an acute inflammatory, demyelinating attack of the optic nerve that triggers neurodegeneration in the entire visual pathway; translating into visual dysfunction. Currently, no neuroprotective therapy with satisfying evidence can be offered to patients. Repetitive transorbital alternating current stimulation (rtACS) is a methodology applied to electrically stimulate the retina and the optic nerve and is considered having neuroprotective- and restorative potential. The goal of this pilot study is to assess safety, tolerability and preliminary efficacy of rtACS as a treatment to improve visual functional as well as structural retinal outcomes in patients with a first-ever episode of autoimmune acute ON.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Informed Consent as documented by signature
* Participants are capable of giving informed consent
* Participant who have a good knowledge of German (patient information and consent must be understood)
* Patients, presenting with typical signs and symptoms suggestive of a first-ever episode of unilateral acute autoimmune, inflammatory, demyelinating ON, including idiopathic ON and ON suggestive of multiple sclerosis (MS) (typical clinically isolated syndrome, or with an established diagnosis of relapsing-remitting MS according to latest panel criteria and no better explanation)
* Patients with high-contrast visual acuity of ≤ 0.63 (decimal system) corresponding to a LogMAR value of ≥ 0.2 on the affected eye (assessed using a Snellen chart during clinical routine)
* Patients presenting in clinics within 14 days of symptom onset
* In principle 18-50 year old female and male patients may be recruited. However, since the randomization of patients will be controlled for gender and participants will be enrolled one at a time on a continuous basis, the gender might become relevant late in the study (e.g. if the female block has already been fully recruited and only males might still be enrolled).
* Patients are receiving standard-of-care treatment for ON (cortisone therapy)

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial
* Women who are pregnant or have the intention to become pregnant during the course of the study (For women who can get pregnant, pregnancy will be omitted using a pregnancy test when checking for inclusion and exclusion criteria. Patients will be informed that they must use contraception during the study)
* Patients with a previous clinical history of ON in the respective eye
* Patients with obvious retinal pathology other than that associated with ON
* Patients who are unable to perform the study assessments (e.g. OCT examination) because of a severe nystagmus (repetitive, uncontrolled eye movements causing unsteady fixation)
* Patients with a recent eye surgery
* Patients with known anti-aquaporin-4- or myelin oligodendrocyte glycoprotein- antibody seropositivity
* Patients with contraindications to the class of device under study (for rtACS): implanted electronic devices, metallic artefacts in the head (excluding dentition), epilepsy, brain cancer, pregnancy, breastfeeding, increased intraocular pressure without appropriate treatment, arterial hypertension without appropriate treatment, skin irritations at intended positions of electrodes, cognitive deficits (unable to provide written informed consent or follow the instructions)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug/device within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — In principle 18-50 year old female and male patients may be recruited. However, since the randomization of patients will be controlled for gender, and participants will be enrolled continuously in an unbiased fashion, gender might become relevant in an advanced phase of the study (e.g. if the female block has already been fully recruited and only males might still be enrolled). As female preponderance is a well-known fact in multiple sclerosis, the investigators anticipate that approximately 2/3 of the patients will be females.
Enrollment: 2 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
The primary functional outcome measure will be low-contrast visual acuity [LogMAR] at 16 weeks (3 month follow-up) in ON eyes. | 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
The primary structural outcome measure will be the mean change in macular ganglion cell and inner plexiform layer thickness [µm] of the affected ON eye at 16 weeks in comparison to baseline of the unaffected contralateral NON eye (pre-treatment). | Baseline (pre-treatment, i.e. 1 week after recruitment), 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
The primary safety outcome measure will be the total number of adverse events during the entire study period | up to 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)

SECONDARY OUTCOMES:
Low-contrast visual acuity [LogMAR] at 4 (post-treatment) weeks in ON eyes. | post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)
The mean change in macular ganglion cell and inner plexiform layer thickness [µm] of the affected ON eye at 4 weeks in comparison to baseline of the unaffected contralateral NON eye (pre-treatment). | Baseline (pre-treatment, i.e. 1 week after recruitment), post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)
High-contrast visual acuity [LogMAR] at 16 weeks (3 month follow-up) in ON eyes. | 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
High-contrast visual acuity [LogMAR] at 4 weeks (post-treatment) in ON eyes. | post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)
Colour vision [tritan] at 16 weeks (3 month follow-up) in ON eyes. | 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
Colour vision [tritan] at 4 weeks (post-treatment) in ON eyes. | post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)
Visual field testing [dB] at 16 weeks (3 month follow-up) in ON eyes. | 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
Visual field testing [dB] at 4 weeks (post-treatment) in ON eyes. | post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)
Recovery of pattern-reversal visual evoked potential conduction velocity of the affected optic nerve [ms] compared to the intra-individual baseline of the unaffected optic nerve at 16 weeks (3 month follow-up). | Baseline (pre-treatment, i.e. 1 week after recruitment), 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
Patient-reported vision-related quality of life assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) at 16 weeks (3 month follow-up). | 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
  The questionnaire contains the following 12 sub-scales: general health, general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, colour vision and peripheral vision. The mean VFQ-25 composite score (calculated as an unweighted average of responses to all items except for the general health sub-scale) and selected sub-scale scores will be analysed. Each sub-scale, and also the composite score, will be quantified with values between 0-100, with zero being the worst and 100 being the best.
Patient-reported vision-related quality of life assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) at 4 weeks (post-treatment). | post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)
  The questionnaire contains the following 12 sub-scales: general health, general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, colour vision and peripheral vision. The mean VFQ-25 composite score (calculated as an unweighted average of responses to all items except for the general health sub-scale) and selected sub-scale scores will be analysed. Each sub-scale, and also the composite score, will be quantified with values between 0-100, with zero being the worst and 100 being the best.
The mean change in peripapillary retinal nerve fibre layer (pRNFL) thickness [µm] of the affected ON eye at 16 weeks (3 month follow-up) in comparison to baseline of the contralateral NON eye. | Baseline (pre-treatment, i.e. 1 week after recruitment), 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
The mean change in peripapillary retinal nerve fibre layer (pRNFL) thickness [µm] of the affected ON eye at 4 weeks (post-treatment) in comparison to baseline of the contralateral NON eye. | Baseline (pre-treatment, i.e. 1 week after recruitment), post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)
The mean change in macular inner nuclear layer (INL) thickness [µm] of the affected ON eye at 16 weeks (3 month follow-up) in comparison to baseline of the contralateral NON eye. | Baseline (pre-treatment, i.e. 1 week after recruitment), 3 month follow-up (16 weeks after recruitment, i.e. 3 months after the last treatment day)
The mean change in macular inner nuclear layer (INL) thickness [µm] of the affected ON eye at 4 (post-treatment) weeks in comparison to baseline of the contralateral NON eye. | Baseline (pre-treatment, i.e. 1 week after recruitment), post-treatment (4 weeks after recruitment, i.e. one week after the last treatment day)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Lutterotti, Prof. Dr. med., Principal Investigator — Neuroimmunology and Multiple Sclerosis Research, Department of Neurology, University Hospital Zurich and University of Zurich, Zurich, Switzerland
Locations (1):
- Department of Neurology and Department of Ophthalmology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No